CLINICAL TRIAL: NCT02640911
Title: An Observational Study on Atypical Antipsychotics Long-term Treatment Patients With Schizophrenia
Status: Recruiting | Type: Observational
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Other Study IDs: SALT-C
Record Dates: First submitted 2015-09-08; First posted 2015-12-29 (Estimated); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This multi-centre study will evaluate the safety and related factors study of atypical antipsychotics long-term treatment in Chinese Patients with Schizophrenia. The atypical antipsychotics include quetiapine, olanzapine, risperidone, aripiprazole, ziprasidone, paliperidone , amisulpride , perospirone and clozapine. This is an open, cohort, multi-center observational clinical study. The main purpose is to evaluate the safety. And the second purpose is to evaluate the efficacy of atypical antipsychotics. The efficacy evaluations include symptoms, social function, recurrence rate and hospitalization. This study belongs to IV period post-marketing drugs research. Planned sample size is 3000 cases.

Visits occurs at 0,4,8,13,26,52,78,104,130 and 156 weeks. The main indexes include physical examination, vital signs, abdominal circumference , laboratory tests (blood cell analysis/ blood biochemical tests / prolactin (PRL) / thyroxine, etc.), adverse events, 12-lead electrocardiogram( ECG), extrapyramidal syndrome(EPS )assessment, sexual function evaluation, medication and other subjective feelings. The second indexes include scales of Positive and Negative Syndrome Scale(PANSS)，Clinical Global Impression-severity of Illness Scale(CGI-S), Calgary Depression Scale for Schizophrenia(CDSS),Personal and Social Performance Scale(PSP), the MOS 36一item Short Form Health Survey(SF-36), relapse rate, drug consolidation, medical-related expenses, income, drug plasma concentration and genetic information.

ELIGIBILITY:
Inclusion Criteria:

1. An in-patient or out-patient (male or female) and aged ≥18 years
2. A diagnosis of schizophrenia,DSM-IV(Diagnostic and Statistical Manual Diploma in Social Medicine-IV)
3. Subjects must have the ability to effectively communicate with investigator,complete study related documents, comprehend the key components of the consent form and must provide written informed consent to participate in the study prior to any study specific assessments or procedures.
4. Patients are taking or will take atypical antipsychotics which include quetiapine, olanzapine, risperidone, aripiprazole, ziprasidone, paliperidone , amisulpride , perospirone and clozapine

Exclusion Criteria:

1. Participation in other clinical studies.
2. Other conditions which, in the investigator's judgment, render patients unsuitable for the clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese Patients with Schizophrenia
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2010-11; Primary Completion 2030-05 (Estimated); Study Completion 2033-05 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Systolic Blood Pressure | at 156 weeks
  Measure blood pressure at 156 weeks
Change from Baseline liver function | at 156 weeks
  Measure blood biochemical tests at 156 weeks
Change from Baseline PRL | at 156 weeks
  Measure PRL level at 156 weeks
Change from Baseline thyroxine | at 156 weeks
  thyroxine laboratory tests at 156 weeks
Number of Participants with EPS | at 156 weeks
  EPS assessment at 156 weeks
Number of Participants with abnormal ECG | at 156 weeks
  ECG examination at 156 weeks
Number of participants with abnormal sexual function | at 156 weeks
  sexual function evaluation medication at 156 weeks

SECONDARY OUTCOMES:
Change from Baseline deduction of PANSS | at 156 weeks
  PANSS assessment at 156 weeks
Change from Baseline deduction of CGI-S | at 156 weeks
  CGI-S assessment at 156 weeks
Change from Baseline deduction of CDSS | at 156 weeks
  CDSS assessment at 156 weeks
Change from Baseline deduction of PSP | at 156 weeks
  PSP assessment at 156 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Weng J, Zhang L, Yu W, Zhao N, Zhu B, Ye C, Zhang Z, Ma C, Li Y, Yu Y, Li H. Risk factors, clinical correlates, and social functions of Chinese schizophrenia patients with drug-induced parkinsonism: A cross-sectional analysis of a multicenter, observational, real-world, prospective cohort study. Front Pharmacol. 2023 Mar 3;14:1077607. doi: 10.3389/fphar.2023.1077607. eCollection 2023. PMID 36937864
- [Derived] He S, Yu WJ, Wang X, Zhang L, Zhao N, Li G, Shen YF, Li H. Risk factors of hyperprolactinemia induced by risperidone and olanzapine and their correlations with plasma glucose and lipids. Gen Psychiatr. 2020 Jul 6;33(4):e100206. doi: 10.1136/gpsych-2020-100206. eCollection 2020. PMID 32695960